CLINICAL TRIAL: NCT03534336
Title: Behavioral Economics-Based Online Lifestyle Balance Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Prof Ho Teck Hua, Professor, National University of Singapore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: A-14-071
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Weight Reduction; Health Knowledge, Attitudes, Practice
Keywords: Weight Reduction; Health Literacy; Financial Incentives; Lifestyle Change
MeSH Terms: conditions — Weight Loss; Behavior | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: 3-arm RCT (Control, Incentive for Weight Loss, Incentive for Education) stratified by Gender.
Who Masked: Participant
Masking Description: A participant knows only the information that is specific to his/her arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants are enrolled in a 12-week, self-administered online weight loss program. The program is delivered through 12 weekly sessions; each includes educational videos and a health literacy quiz. Each quiz contains 10 questions, and a quiz is considered "passed" when at least 7 questions are answered correctly. All participants are encouraged to follow the program, take the quizzes, and lose 5% of their baseline body weight by the end of the program.
  No financial incentives are given for losing weight or passing quizzes.
- Incentive for Education (Experimental): Same 12-week, self-administered online weight loss program as in the Control arm.
  Each participant is also given a $150 "Incentive for Education" for passing at least nine quizzes by the end of the program.
  Interventions: Behavioral: Incentive for Education
- Incentive for Weight Loss (Experimental): Same 12-week, self-administered online weight loss program as in the Control arm.
  Each participant is also given a $150 "Incentive for Weight Loss" for losing 5% of their baseline body weight.
  Interventions: Behavioral: Incentive for Weight Loss

INTERVENTIONS:
Behavioral: Incentive for Education — A $150 "Incentive for Education" is given to the participants for passing at least nine quizzes by the end of the program
  Arms: Incentive for Education
Behavioral: Incentive for Weight Loss — A $150 "Incentive for Weight Loss" is given to the participants for losing at least 5% of baseline weight by the end of the program
  Arms: Incentive for Weight Loss

SUMMARY:
The objective of this project is to design a Behavioral Economics Based Online Lifestyle Balance Program that employs behavioral economics to engage and motivate adherence to an Internet-based program. The investigators compare the effects of two financial incentives on inducing weight loss: a direct financial incentive for weight loss and a financial incentive for health literacy.

DETAILED DESCRIPTION:
This project investigates whether participants in an online weight loss program can be induced to achieve weight loss using financial incentives. The study is a 3-arm randomized controlled trial (RCT) stratified by gender. The goal is to examine how overweight individuals respond to two different types of financial incentives. The first type of incentive, incentive for weight loss (IW), is a cash award of approximately $150 given for achieving 5% weight loss over 12 weeks. The second type of incentive, incentive for education (IE), is a $150 award for passing quizzes that test the participants' health literacy about weight loss and the techniques required for maintaining a healthy lifestyle. The investigators compare the effectiveness of IW to IE in promoting weight loss in overweight individuals and investigate whether the two incentives work equally well for men and women.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 23 and 33
* Age between 40 and 60 years old

Exclusion Criteria:

* History of diabetes
* History of significant cardiovascular disease
* Family history of atherosclerosis
* High blood pressure
* Significant lung disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 710 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-06-22 (Actual)

PRIMARY OUTCOMES:
Weight Loss at the end of the weight loss program (at Week 13) | At week 13 of the RCT.
  Weight measured at the Week 13 weigh-in session. Weight measurements are taken by trained research assistants using digital scales.

SECONDARY OUTCOMES:
Weight Loss at the end of the post-intervention period (Week 25) | At week 25 of the RCT.
  Weight measured at the Week 25 weigh-in session. Weight measurements are taken by trained research assistants using digital scales.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the research, after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.